CLINICAL TRIAL: NCT07357246
Title: The Effect of Breathing Exercises Applied Under the Guidance of Student Midwives During Birth on Labor Pain, Labor Duration and Birth Satisfaction: A Randomized Controlled Trial
Brief Title: Breathing Exercises Guided by Student Midwives During Labor
Acronym: BREATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Bilim University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2026-SS; 1919B012324751 (Other Grant/Funding Number: TUBITAK 2209-A Undergraduate Research Support Program)
Record Dates: First submitted 2026-01-02; First posted 2026-01-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Labor Pain and to Reduce Pain; Childbirth; Normal Labor
Keywords: Breathing Exercises; Labor Pain; Student Midwives; Birth Satisfaction; Labor Duration; Midwifery Care
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercises Guided by Student Midwives (Experimental): Participants in this group will receive structured breathing exercises in addition to routine intrapartum care. The breathing exercises will be guided by trained student midwives from admission to the labor ward until birth. The intervention will include slow-paced breathing, patterned breathing during contractions, and relaxation-focused breathing between contractions, with continuous guidance and encouragement provided according to a standardized protocol.
  Interventions: Behavioral: Guided Breathing Exercises During Labor
- Routine Intrapartum Care (Active Comparator): Participants in this group will receive routine intrapartum care according to the standard clinical protocols of the maternity hospital. Routine care includes regular maternal and fetal monitoring, clinical assessment by midwives and obstetric staff, support during labor as per standard practice, and medical or obstetric interventions if clinically indicated. No structured breathing exercise program will be provided.
  Interventions: Other: Routine Intrapartum Care

INTERVENTIONS:
Behavioral: Guided Breathing Exercises During Labor — Structured breathing exercises delivered and monitored by student midwives during labor.
  Arms: Breathing Exercises Guided by Student Midwives
Other: Routine Intrapartum Care — Standard intrapartum care provided according to hospital protocols.
  Arms: Routine Intrapartum Care

SUMMARY:
This randomized controlled trial aimed to evaluate the effect of breathing exercises applied under the guidance of student midwives during labor on labor pain, labor duration, and birth satisfaction. The intervention group received structured breathing exercises guided by student midwives throughout labor, while the control group received routine intrapartum care. Outcomes were assessed during labor and in the early postpartum period

DETAILED DESCRIPTION:
This study is designed to evaluate the effect of a midwifery-led intervention on labor pain intensity and birth satisfaction among women giving birth vaginally. The study will be conducted as a controlled clinical study in a maternity hospital setting. Eligible pregnant women who are admitted to the labor ward and meet the inclusion criteria will be invited to participate and will provide informed consent prior to enrollment.

The study aims to determine whether the midwifery-led intervention is associated with reduced labor pain intensity and improved birth satisfaction compared to routine care.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older

Term pregnancy (≥37 weeks of gestation)

Singleton pregnancy

Planning vaginal birth

In the active phase of labor

Able to communicate and provide informed consent

Exclusion Criteria:

* High-risk pregnancy (e.g., preeclampsia, placenta previa, severe medical complications)

Multiple pregnancy

Planned cesarean section

Use of pharmacological pain relief at admission (e.g., epidural analgesia)

Known fetal anomalies

Inability to participate in breathing exercises

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Labor pain intensity measured by the Visual Analog Scale (VAS) (0-10) | At admission to the labor ward (baseline) and at cervical dilatation of 6-7 cm.
  Labor pain intensity will be assessed using a 10-cm Visual Analog Scale (VAS), where 0 indicates "no pain" and 10 indicates "worst pain imaginable." The outcome will be the VAS score reported by the participant at each assessment time point.

SECONDARY OUTCOMES:
Birth satisfaction measured by the Birth Satisfaction Scale Revised (BSS-R) | Within the first 24 hours postpartum
  Birth satisfaction will be assessed using the Birth Satisfaction Scale-Revised (BSS-R), a 10-item scale with total scores ranging from 0 to 40, where higher scores indicate greater birth satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Serhatlioglu, Doctorate, Principal Investigator — Antalya Bilim Üniversitesi
Locations (1):
- Antalya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared.